CLINICAL TRIAL: NCT05895656
Title: Exploration of Knee Injuries Using 3 Tesla and 7 Tesla Magnetic Resonance Imaging at the University Hospital of Poitiers.
Acronym: MR7T-KneeTraum
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MR7T-KneeTraumatic
Record Dates: First submitted 2023-05-22; First posted 2023-06-08 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Traumatic Knee Injury; Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 7 Tesla MRI — Performing an additional 7 Tesla MRI examination as part of the initial treatment pathway.

SUMMARY:
The knee is the most stressed and exposed joint in sports practice (70 to 85% of Anterior Cruciate Ligament ruptures occur during sports activities). Although traumatic knee injuries are already described in radiology and 1.5 Tesla and 3 Tesla MRI, there are cases of post-traumatic knee pain with a normal MRI (with a risk of underestimating a traumatic injury that may worsen without appropriate treatment) and cases of "ambiguous" MRI findings (uncertainty between low or high-grade ligament or meniscal injury, presence or absence of meniscal attachments, complete versus partial rupture of the Anterior Cruciate Ligament, associated cartilage lesion versus intact cartilage), which directly impact orthopedic or surgical therapeutic management.

DETAILED DESCRIPTION:
Knee pain (or gonalgia) is a very common complaint in the general population, accounting for nearly 6% of visits to general practitioners and experienced by approximately 46% of patients at least once in their lifetime (Jackson et al.).

The knee is one of the largest and most complex joints in the body, comprising three different joints and a multitude of stabilizing and functional structures (ligaments, menisci, bursa, tendons, etc.).

This complex functional anatomy partly explains the multiple etiologies of knee pain, especially post-traumatic. Among these etiologies, ligamentous (particularly anterior cruciate ligament), bony, and meniscal injuries are prominent (Webb et al.).

The passive stability of the knee is ensured by a complex capsuloligamentary system. Two ligament systems are usually distinguished: the central pivot (cruciate ligaments) and the peripheral structures (anterior, anterolateral, collateral, and posterior). In the case of injuries to one or more elements of this system, knee instability can occur and be detrimental to functional prognosis. These injuries should be addressed promptly (Bressy et al.).

Furthermore, these capsuloligamentary injuries are frequently associated with complex meniscal, bony, or musculotendinous lesions (Blin et al., Boutry et al.).

With surgical techniques becoming increasingly precise and minimally invasive, surgeons need accurate preoperative localization of these lesions to plan their surgical approach and operative procedure (Fanelli - book).

These injuries are better understood with 3 Tesla MRI, which is the imaging modality of choice, in addition to standard radiographs, for exploring traumatic knee injuries (Blin et al.). MRI, by visualizing contusion areas, helps understand the mechanism of trauma and predict and confirm capsuloligamentary injuries.

However, in our clinical practice, we observe that a certain percentage of MRI examinations are considered unremarkable despite patients experiencing persistent post-traumatic pain or functional discomfort. This could be related to insufficient imaging resolution in relation to the millimetric nature of the explored lesions.

Considering all this data, it has become pertinent for us to:

* Seek to optimize the diagnostic quality of MRI imaging in these patients, as it directly affects orthopedic management.
* Seek to improve existing MRI lesion classifications and develop new ones.
* Develop new MRI tools (sequences) for exploring traumatic knee injuries.

The expected results are:

* Define the 7 Tesla MRI findings of traumatic knee injuries.
* Assess the inter-observer variability between 3T and 7T for a future study on diagnostic power (preliminary data).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 60 years
* Knee injury less than 2 months old
* Patients who have undergone or will undergo a 3T MRI
* Subject with no contraindication to MRI (metallic splinter, pacemaker, …)
* Free subject, without guardianship or curatorship or subordination
* Patient benefiting from a Social Security plan or benefiting from it through a third through a third party
* Informed consent signed by the patient after clear and fair information on the study

Exclusion Criteria:

* Subjects with contraindications to 7T MRI (pregnancy, metallic fragments, pacemakers, copper intrauterine devices, tattoos larger than 5 cm in examination area, stents, coils, ocular metallic foreign bodies (accidental or otherwise), cochlear implants, and generally any electronically implanted medical device; metallic heart valves, previously implanted vascular clips on a cranial aneurysm)
* History of knee surgery.
* Patient without Social Security coverage or coverage through a third party.
* Patient suffering from claustrophobia.
* Individuals benefiting from enhanced protection, namely minors, persons deprived of liberty by a judicial or administrative decision, adults under legal protection, and emergency patients.
* Pregnant or breastfeeding women, women of childbearing age without effective contraception (hormonal/mechanical: oral, injectable, transdermal, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Describe and quantify post-traumatic injuries of the ligaments (Anterior Cruciate Ligament, Posterior Cruciate Ligament, Lateral Collateral Ligament, Medial Collateral Ligament) using 7T MRI compared to 3T MRI in cases of post-traumatic knee pain. | 27 to 30 months
  For the Anterior Cruciate Ligament (ACL) and Posterior Cruciate Ligament (PCL), they will be described and classified as follows: no abnormality, complete rupture, or partial rupture depending on the location (proximal, medial, distal). For the Lateral Collateral Ligament (LCL) and Medial Collateral Ligament (MCL), the ligament classification will be applied (3 grades).

SECONDARY OUTCOMES:
Describe and quantify post-traumatic meniscal injuries using 7T MRI compared to 3T MRI in cases of post-traumatic knee pain. | 27 to 30 months
  For the menisci, the classification of Israkes, Trillat, Arnoczky, and Warren will be applied.
Describe and quantify post-traumatic musculotendinous injuries using 7T MRI compared to 3T MRI in cases of post-traumatic knee pain. | 27 to 30 months
  For musculoskeletal injuries:
  - 3 grades will be used: inflammatory, partial rupture, complete rupture.
Describe and quantify post-traumatic bone injuries using 7T MRI compared to 3T MRI in cases of post-traumatic knee pain. | 27 to 30 months
  For bone injuries:
  - 3 grades will be used: bone edema, subchondral fissure, fracture.
Describe and quantify post-traumatic cartilage injuries using 7T MRI compared to 3T MRI in cases of post-traumatic knee pain. | 27 to 30 months
  For cartilage injuries, the Outerbridge classification will be applied.
Evaluate Cohen's Kappa coefficient value to quantify the inter-rater reliability with 3 and 7 Tesla MRI findings | 27 to 30 months
  The inter- and intra-observer study will be conducted by reviewing the images by different radiologists. This will allow us to quantify the variability by comparing the assessment criteria.
Evaluate Cohen's Kappa coefficient value to quantify the intra-rater reliability with 3 and 7 Tesla MRI findings | 27 to 30 months
  The inter- and intra-observer study will be conducted by reviewing the images by different radiologists. This will allow us to quantify the variability by comparing the assessment criteria.
Compare the 7T structural MRI findings of traumatic knee injuries to the structural findings of the surgical reports | 27 to 30 months
  For defining the semiotics, the MRI report at 7T will be compared to the surgical report, if applicable. The surgical report will be considered as the reference for the lesions identified by the surgeon (as arthroscopy is the gold standard examination).